CLINICAL TRIAL: NCT07321561
Title: The Effect of Motor Support Program Applıed to Chıldren wıth Autısm Spectrum Dısorder on Gross Motor and Sensory Motor
Brief Title: Effect of a Motor Support Program in Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gökçe Oktay, Assistant Professor, Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IUC-SBBEK-2024-143
Record Dates: First submitted 2025-12-19; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Motor Skil; Sensory motor skill; Motor Support Program
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: A total of 28 children with ASD participated in the study, 14 students in the experimental group and 14 in the control group. In addition to the special education sessions, the participants in the experimental group received a motor support program for 40 minutes 2 days a week for 12 weeks. In the study, the Gilliam Autistic Disorder Rating Scale-2-TV, the Bruininks-Oseretsky Motor Competence 2 Test Short Form (BOT-2) for the assessment of gross motor skills, and the caregiver sensory profile questionnaire for the assessment of sensory-motor skills were used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Support Program (Experimental): The motor support program (MSP) consists of activities prepared by the researchers by taking into account the test protocols used to achieve desired changes in children's gross motor (throwing, jumping, catching, running, etc.), sensory-motor (sensory modulation, sensory processing, sensory inputs related to movement) skill levels and developmental areas.
  Interventions: Other: Motor Support Program
- Standard Education (No Motor Support) (No Intervention): Participants in the control group continued their individual education programs. However, they did not participate in any physiotherapy or motor support programs. Only pre- and post-test measurements were taken.

INTERVENTIONS:
Other: Motor Support Program — The MSP was administered by the first researcher for 60 minutes, 2 days a week for 12 weeks at the special education center where they were studying. A special program was prepared for the first 10 weeks, and in the last 2 weeks, a choose your activity activity was conducted. During this activity, children were presented with different options consisting of the activities implemented in the first 8 weeks and were asked to choose and implement them. Within each lesson plan, at least 3 different game formats were implemented for children's gross motor skills and sensory motor skills. In the following weeks, different game formats aime
  Arms: Motor Support Program

SUMMARY:
This study examined a motor support program applied for 40 minutes, two days per week, over a period of 12 weeks in children aged 4-6 years diagnosed with autism spectrum disorder. A total of 28 children with autism spectrum disorder participated in the study, including 14 children in the experimental group and 14 children in the control group. In addition to their regular special education sessions, participants in the experimental group received the motor support program for 40 minutes, two days per week, for 12 weeks. Data collection instruments included the Gilliam Autistic Disorder Rating Scale-Second Edition, Turkish Version (GARS-2-TV), the Bruininks-Oseretsky Test of Motor Proficiency, Second Edition, Short Form (BOT-2) for the assessment of gross motor skills, and the caregiver-completed Sensory Profile Questionnaire for the assessment of sensory-motor skills.

DETAILED DESCRIPTION:
This study is a quasi-experimental research design including pretest-posttest experimental and control groups, and one of the previously determined groups was randomly assigned as the experimental group and the other as the control group. The study was conducted with a total of 28 children, including 14 children in the control group (CG) and 14 children in the experimental group (EG), aged between 4 and 6 years, diagnosed with autism spectrum disorder, who were continuing their education in special education and rehabilitation centers located in the Bayrampaşa and Esenyurt districts of Istanbul. The number of participants was determined using G*Power analysis, with a statistical power of 0.80, an effect size of 0.05, and a margin of error of 0.05. The inclusion criteria were defined as being between the ages of 4 and 6 years, having a diagnosis of autism spectrum disorder, having no additional intellectual disability, and having no health condition that would prevent participation in physical activity. Data collection instruments included the Gilliam Autistic Disorder Rating Scale-Second Edition, Turkish Version (GARS-2-TV), the Bruininks-Oseretsky Test of Motor Proficiency, Second Edition, Short Form (BOT-2) for the assessment of gross motor skills, and the caregiver-completed Sensory Profile Questionnaire for the assessment of sensory-motor skills. The BOT-2 Short Form was administered in approximately 20-25 minutes per child. The GARS-2-TV, administered through interviews with caregivers, was completed in approximately 25-30 minutes per child. The Sensory Profile Questionnaire was completed by caregivers in approximately 30-35 minutes per child. As the GARS-2-TV requires certification for administration, the required training and certification were obtained by the evaluator.The motor support program (MSP) consisted of activities prepared in accordance with test protocols to support children's gross motor skills (e.g., throwing, jumping, catching, running) and sensory-motor skills (e.g., sensory modulation, sensory processing, and movement-related sensory input). The MSP was implemented for 60 minutes per session, two days per week, over a period of 12 weeks at the special education centers attended by the participants. A structured program was applied during the first 10 weeks, and during the final 2 weeks, a "choose-your-activity" approach was implemented, in which children selected activities from those applied during the previous weeks. Within each session, at least three different game-based activity formats targeting gross motor and sensory-motor skills were implemented. In subsequent weeks, different game formats were included to address multiple developmental domains.

ELIGIBILITY:
Inclusion Criteria:

* Being between 4 and 6 years of age
* Having no health problems that would prevent participation in the study
* Having been diagnosed with autism according to the Health Board and Guidance and Research Center (RAM) report
* Not having previously participated in any motor-supported education programs (e.g., occupational therapy sessions)
* Having no additional diagnoses related to physical or intellectual disabilities other than autism spectrum disorder

Exclusion Criteria:

* The participant's failure to attend the training program for three consecutive sessions
* The participant's failure to fulfill the assigned responsibilities
* The participant's voluntary withdrawal from the study at any stage for any reason

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Change in Motor Skills as Measured by the Bruininks-Oseretsky Test of Motor Proficiency, Second Edition - Short Form (BOT-2 SF)" | Evaluations were conducted at three time points: at baseline (pretest), at the end of the 12-week intervention (posttest).
  In this study, the short form of the Bruininks-Oseretsky Motor Competence Test-2 (BOT-2 SF), which was developed to assess the motor skill levels of individuals aged 4-21 years, was used. The short form used in the study consists of a total of eight subtests and 12 items. These subtests include fine motor accuracy, fine motor integration, manual agility, two-way coordination, balance, running speed and agility, hand-arm coordination and strength. The maximum score that can be obtained in the test is 50. As the total score increases, the level of motor skills increases.
Sensory profile questionnaire to assess sensory motor skills | Evaluations were conducted at three time points: at baseline (pretest), at the end of the 12-week intervention (posttest).
  The Sensory Profile Scala was designed by Dunn in 1999 to assess children's sensory processing skills and is administered to children aged 3-10 years. The scale aims to assess the sensory reactions of children in their daily lives and is completed by the caregiver. Turkish adaptation, validity and reliability study was conducted by Kayıhan et al. The Sensory Profile Scale consists of three main sections and their sub-sections: (1) Sensory processing, (2) Sensory modulation, and (3) Behavioral-emotional responses. The scale, which consists of 125 items in total, is structured to assess the frequency of children's behaviors in response to different sensory stimuli. The items are scored on a 5-point Likert-type rating system. In this system, "Always" response is evaluated as 1 point and "Never" response is evaluated as 5 points.As the total score on the scale increases, sensory regulation skills improve.
The Gilliam Autism Rating Scale-2 (GADRS) for the assessment of autism-related symptoms. | Evaluations were conducted at three time points: at baseline (pretest), at the end of the 12-week intervention (posttest).
  This scale was developed by Gilliam (2006) to diagnose children with autism spectrum disorder. The scale is completed by caregivers. The scale consists of 3 sub-dimensions."0" means never observed while '3' means frequently observed. The scale consists of 42 items. The highest standard score that can be obtained from this scale is 153, and the lowest score is 55. A high total score indicates a high probability of ASD. A low score indicates a low likelihood of ASD. Since the Gilliam Autistic Disorder Rating Scale-2 is a scale that can be used with a certificate, the necessary training and certificate were obtained by the researcher.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydin University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bruininks RH, & Oseretsky, B. D., 2010, Bruininks-Oseretsky Test Of Motor Proficiency, Second Edition, Brief Form. Bloomington: Psychcorp.
- [Background] Kayıhan H, Günel M. K, Bumin G. Adaptation of the Sensory Profile into Turkish for children aged 3-10 years: A validity and reliability study. Turkish Journal of Physiotherapy and Rehabilitation. 2011; 22(2): 44-53.